CLINICAL TRIAL: NCT00329888
Title: Comparison of Endoscopic Papillary Balloon Dilatation and Sphincterotomy for CBD Stones With Difficult Sphincterotomy or Distal CBD Tapering
Brief Title: Comparison of Papillary Balloon Dilatation Vs.Sphincterotomy for Lithotripsy in Difficult Sphincterotomy or Distal CBD Tapering
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9561703024
Record Dates: First submitted 2006-05-24; First posted 2006-05-25 (Estimated); Last update posted 2006-05-25 (Estimated); Status verified 2006-04

CONDITIONS: Choledocholithiasis
Keywords: Endoscopic papillary balloon dilatation; Endoscopic sphincterotomy
MeSH Terms: conditions — Choledocholithiasis | interventions — Sphincterotomy, Endoscopic

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Procedure: Endoscopic papillary balloon dilatation
Procedure: Endoscopic sphincterotomy

SUMMARY:
Compare endoscopic papillary balloon dilatation vs. endoscopic sphincterotomy for bile duct stones in:

* when sphincterotomy is difficult (periampullary diverticulum, prior sphincterotomy or Billroth II anastomosis)
* when there is distal CBD tapering.

DETAILED DESCRIPTION:
Endoscopic papillary balloon dilatation is an alternative to endoscopic sphincterotomy for treating bile duct stones:

* easier and as effective. But...
* a higher risk of pancreatitis.

Conditions including periampullary diverticulum, prior EST, Billroth-II anastomosis, or distal CBD tapering pose difficulty in EST and lithotripsy with increased risk of complications.

Whether EPBD or EST is superior in efficacy or safety under such circumstances is not clear.

ELIGIBILITY:
Inclusion Criteria:

* Choledocholithiasis with
* Difficult sphincterotomy:periampullary diverticulum, prior sphincterotomy or Billroth II anastomosis
* or distal CBD tapering.

Exclusion Criteria:

* Patients in whom no endoscopic papillary balloon dilatation or endoscopic sphincterotomy was performed for lithotripsy

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2006-03; Study Completion 2006-05

CONTACTS AND LOCATIONS:
Overall Officials: Wei Chih Liao, MD., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] 1. Minami A, Nakatsu T, Uchida N, Hirabayashi S, Fukuma H, Morshed SA, Nishioka M. Papillary dilation vs sphincterotomy in endoscopic removal of bile duct stones. A randomized trial with manometric function. Dig Dis Sci 1995;40:2550-4. 2. Bergman JJ, Rauws EA, Fockens P, van Berkel AM, Bossuyt PM, Tijssen JG, Tytgat GN, Huibregtse K. Randomised trial of endoscopic balloon dilation versus endoscopic sphincterotomy for removal of bile duct stones. Lancet 1997;349:1124-9. 3.Komatsu Y, Kawabe T, Toda N, Ohashi M, Isayama M, Tateishi K, Sato S, Koike Y, Yamagata M, Tada M, Shiratori Y, Yamada H, Ihori M, Kawase T, Omata M. Endoscopic papillary balloon dilation for the management of common bile duct stones: experience of 226 cases. Endoscopy 1998;30:12-7. 4. Fujita N, Maguchi H, Komatsu Y, Yasuda I, Hasebe O, Igarashi Y, Murakami A, Mukai H, Fujii T, Yamao K, Maeshiro K. Endoscopic sphincterotomy and endoscopic papillary balloon dilatation for bile duct stones: A prospective randomized controlled multicenter trial. Gastrointest Endosc 2003;57:151-5.